CLINICAL TRIAL: NCT01149824
Title: A Double Blind Placebo Controlled Ascending Dose Pharmacodynamic and Tolerability Study of 100 to 4000 µg of Sublingual Salvinorin A
Brief Title: Placebo Controlled Study of Sublingual Salvinorin A
Acronym: 6A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Principal Investigator, John Mendelson, MD, Senior Scientist, California Pacific Medical Center Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: CPMC-APRL-6A
Record Dates: First submitted 2010-06-22; First posted 2010-06-24 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Pharmaceutical Preparations
Keywords: Salvia divinorum; Salvinorin A
MeSH Terms: interventions — salvinorin A

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Dose Escalating (Other)
  Interventions: Drug: Salvinorin A; Drug: Placebo

INTERVENTIONS:
Drug: Salvinorin A
Drug: Placebo

SUMMARY:
In this study, our aim is to determine an active but tolerable sublingual dose (range 100 to 4000 µg) of Salvinorin A (SA) in experienced subjects. This study is an ascending-dose, placebo-controlled, single-site design in 8 Salvia-experienced subjects. Subjects will receive SA doses from 0-4000 µg. Doses will be separated by at least one day. The first two doses (0 and 100µg) will be double-blinded while the last four (250, 500, 1000, 2000 and 4000µg) will be single-blind.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 21-45
* Experienced with hallucinogenic amounts of SA
* Good physical and mental health
* Able to give adequate informed consent

Exclusion Criteria:

* Any medical or psychiatric condition which, in the investigators' opinion, would preclude safe or consistent participation
* Significant acute or chronic medical disease
* Female who is pregnant, lactating, or plans to become pregnant during the study period and within one month after study drug administration

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To determine an active but tolerable sublingual dose (range 100 to 4000 µg) of Salvinorin A (SA) in experienced subjects. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: John Mendelson, MD, Principal Investigator — California Pacific Medical Center